CLINICAL TRIAL: NCT00137969
Title: Randomized, Double-blind, Placebo-controlled, Multicenter, Phase II/III Study to Evaluate the Efficacy and Safety of Rituximab in Subjects With Moderate to Severe Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety of Rituximab Retreatment in Subjects With Systemic Lupus Erythematosus
Acronym: EXPLORER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U2971g
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2017-06

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Rituxan; SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Rituximab; Prednisone; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab 1000 mg + prednisone (Experimental): Participants will receive rituximab 1000 mg intravenously on Days 1, 15, 168, and 182. Participants will also receive an initial dose of prednisone (0.5, 0.75, or 1.0 mg/kg orally once a day) with tapering beginning at Day 16 for 10 weeks to a dose of ≤ 10 mg/day. Participants will also receive acetaminophen 1000 mg orally and diphenhydramine 50 mg orally prior to study drug infusion.
  Interventions: Drug: Rituximab; Drug: Prednisone; Drug: Acetaminophen; Drug: Diphenhydramine
- Placebo + prednisone (Placebo Comparator): Participants will receive placebo intravenously on Days 1, 15, 168, and 182. Participants will also receive an initial dose of prednisone (0.5, 0.75, or 1.0 mg/kg orally once a day) with tapering beginning at Day 16 for 10 weeks to a dose of ≤ 10 mg/day. Participants will also receive acetaminophen 1000 mg orally and diphenhydramine 50 mg orally prior to study drug infusion.
  Interventions: Drug: Placebo; Drug: Prednisone; Drug: Acetaminophen; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Rituximab — Rituximab will be supplied as a sterile liquid for IV administration.
  Other Names: Rituxan; MabThera; Zytux
  Arms: Rituximab 1000 mg + prednisone
Drug: Placebo — Placebo will be supplied as a sterile liquid for IV administration.
  Arms: Placebo + prednisone
Drug: Prednisone
Drug: Acetaminophen
Drug: Diphenhydramine

SUMMARY:
This is a Phase II/III, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of rituximab compared with placebo when combined with a single stable background immunosuppressive medication in subjects with moderate to severe systemic lupus erythematosus (SLE). The primary efficacy endpoint of the trial will be evaluated at 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus (SLE).
* Active disease at screening.
* Stable use of one immunosuppressive drug.
* Use of an antimalarial drug.
* For subjects of reproductive potential (males and females), use of a reliable means of contraception throughout their study participation.

Exclusion Criteria:

* Unstable patients with thrombocytopenia experiencing or at high risk for developing clinically significant bleeding or organ dysfunction requiring therapies such as plasmapheresis or acute blood or platelet transfusions.
* Active moderate to severe glomerulonephritis.
* Retinitis, poorly controlled seizure disorder, acute confusional state, myelitis, stroke or stroke syndrome, cerebellar ataxia, or dementia that is currently active and resulting from SLE.
* Lack of peripheral venous access.
* Pregnant women or nursing (breast feeding) mothers.
* History of severe, allergic, or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Significant, uncontrolled medical disease in any organ system not related to SLE that in the investigator's opinion would preclude subject participation.
* Concomitant conditions that require oral or systemic corticosteroid use.
* Known human immunodeficiency virus (HIV) infection.
* Known active infection of any kind (excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics.
* History of deep space infection.
* History of serious recurrent or chronic infection.
* History of cancer, including solid tumors, hematological malignancies, and carcinoma in situ.
* Active alcohol or drug abuse, or history of alcohol or drug abuse.
* Major surgery.
* Previous treatment with CAMPATH-1H antibody.
* Previous treatment with any B cell-targeted therapy.
* Treatment with any investigational agent within 28 days of screening (Day -7) or 5 half-lives of the investigational drug (whichever is longer).
* Receipt of a live vaccine within 28 days prior to screening.
* Intolerance or contraindication to oral or IV corticosteroids.
* Use of a new immunosuppressive drug prior to screening or change in dose of ongoing immunosuppressive drug prior to screening.
* Prednisone dose of ≥ 1 mg/kg/day prior to screening.
* Treatment with cyclophosphamide or a calcineurin inhibitor.
* Treatment with a second immunosuppressive or immunomodulatory drug.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x the upper limit of normal.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2005-05-10 (Actual); Primary Completion 2008-08-25 (Actual); Study Completion 2008-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Brunetta, M.D., Study Director — Genentech, Inc.
Locations (65):
- United States (63):
  - Univ of Alabama School of Med; Clinical Immun Rheumatology, Birmingham, Alabama
  - Rheumatology Assoc of North AL, Huntsville, Alabama
  - Arizona Arthritis & Rheumatology Research, Pllc, Paradise Valley, Arizona
  - Univ of California, San Diego, La Jolla, California
  - Univ of Calif., Los Angeles; Rheumatology, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Med Ctr;Div of Immunology/Rheumatology, Palo Alto, California
  - Univ of Calif, San Francisco; Rheumatology, San Francisco, California
  - Eden Medical Center San Leandro Hospital, San Leandro, California
  - University of Colorado Denver, Aurora, Colorado
  - Arthritis & Rheumatism; Disease Specialities, Aventura, Florida
  - Family Arthritis Center, Jupiter, Florida
  - Emory Uni ; Division of Rheumatology, Atlanta, Georgia
  - Intermountain Research Center, Boise, Idaho
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Northwestern University, Chicago, Illinois
  - Rheumatology Associates, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tri-State Arth & Rheum Center, Evansville, Indiana
  - Univ of Kansas Medical Center; Allergy/Clin Imm/Rheum, Kansas City, Kansas
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - LA State Univ; Medicine, Shreveport, Louisiana
  - Johns Hopkins Uni, Baltimore, Maryland
  - Center For Rheumatology & Bone Research, Wheaton, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute; Rheumatology, Boston, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Michigan Arthritis Rsrch Ctr, Brighton, Michigan
  - Washington University; Rheumatology Division, St Louis, Missouri
  - Center for Rheumatology, State Uni. of New York, Albany, New York
  - SUNY Downstate Medical Center., Brooklyn, New York
  - NS-LIJ Health Systems; Rheum-Allergy Clin Immu, Lake Success, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - NYU-Hosp for Joint Diseases; Rheum and Med, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Buffalo Rheumatology Associates, Orchard Park, New York
  - Long Island Osteo/Arth Center, Plainview, New York
  - University of Rochester - Strong Memorial Hospital, Rochester, New York
  - University of North Carolina Hospitals Department of Pharmacy; Investigational Drug Services, Chapel Hill, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - Physicians East Pa, Greenville, North Carolina
  - Ohio State University; Division of Nephrology, Columbus, Ohio
  - Bone and Joint Hospital at St. Anthony Research Department, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma Center For Arthritis Therapy & Research, Tulsa, Oklahoma
  - Portland Medical Associates, Portland, Oregon
  - East Penn Rheumatology Associates, Pc, Bethlehem, Pennsylvania
  - Altoona Arthritis & Osteo Center, Duncansville, Pennsylvania
  - Uni of Pennslyvania Medical Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical Univ of South Carolina, Charleston, South Carolina
  - Arthritis Associates PLLC, Chattanooga, Tennessee
  - Metroplex Clinical Research, Dallas, Texas
  - Arthritis Centers of Texas, Dallas, Texas
  - Houston Inst. For Clinical Research, Houston, Texas
  - Arthritis & Osteoporosis Associates, LLP, Lubbock, Texas
  - Texas Research Center, Sugar Land, Texas
  - University of Virginia Med Ctr; Div of Ped Respiratory Med, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Rheumatology Assoc; Swedish Rheumatology Research, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Arthritis Northwest, Spokane, Spokane, Washington
- Canada (2):
  - Univ of Manitoba, Health Scien; Arthritis Centre, Winnipeg, Manitoba
  - St. Joseph'S Health Care Centre, London, Ontario

REFERENCES:
- [Derived] Merrill JT, Neuwelt CM, Wallace DJ, Shanahan JC, Latinis KM, Oates JC, Utset TO, Gordon C, Isenberg DA, Hsieh HJ, Zhang D, Brunetta PG. Efficacy and safety of rituximab in moderately-to-severely active systemic lupus erythematosus: the randomized, double-blind, phase II/III systemic lupus erythematosus evaluation of rituximab trial. Arthritis Rheum. 2010 Jan;62(1):222-33. doi: 10.1002/art.27233. PMID 20039413

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab 1000 mg + Prednisone: Participants received rituximab 1000 mg intravenously (IV) on Days 1, 15, 168, and 182. Participants also received an initial dose of prednisone (0.5, 0.75, or 1.0 mg/kg orally once a day) with tapering beginning at Day 16 for 10 weeks to a dose of ≤ 10 mg/day. Participants also received acetaminophen 1000 mg orally and diphenhydramine 50 mg orally prior to study drug infusion.
- Placebo + Prednisone: Participants received placebo intravenously on Days 1, 15, 168, and 182. Participants also received an initial dose of prednisone (0.5, 0.75, or 1.0 mg/kg orally once a day) with tapering beginning at Day 16 for 10 weeks to a dose of ≤ 10 mg/day. Participants also received acetaminophen 1000 mg orally and diphenhydramine 50 mg orally prior to study drug infusion.
Period: Overall Study
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Started | 174 | 88
Received Study Drug | 169 | 88
Completed | 107 | 67
Not Completed | 67 | 21

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone | Total
Number analyzed (Participants) | 169 | 88 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.4) | 40.5 (12.8) | 40.3 (11.9)
Age, Customized [Number; unit: participants]
  < 20 years | 2 | 2 | 4
  20 to 64 years | 166 | 83 | 249
  > 64 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 82 | 234
  Male | 17 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Major Clinical Response (MCR), Partial Clinical Response (PCR), or Nonclinical Response (NCR) Defined by British Isles Lupus Assessment Group (BILAG) Scores Over The 52-week Treatment Period
Description: The BILAG Index measures clinical disease activity in Systemic Lupus Erythematosus (SLE). A single alphabetic score (A through E) is used to denote disease severity for each of the 8 domains. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 8 domains. MCR = participants who achieved BILAG C scores or better at 24 weeks, maintained this response without developing a flare to 52 weeks, and did not experience a severe flare from Day 1 to Week 24; PCR = participants who achieved BILAG C score or better at 24 wks and maintained response without a flare for 16 consecutive weeks, or maximum of one BILAG B score at 24 weeks and maintained response without a flare to 52 wks, or maximum of 2 BILAG B scores at 24 wks without development of BILAG scores of A or B until Week 52 if the baseline BILAG score was 1A+>=2Bs, or>=2 As, or>=4 Bs, or participants who enrolled with scores of severe disease and did not achieve a single BILAG B at Month 6.
Time Frame: From baseline to 52 weeks
Population: Intent-to-treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 169 | 88
Participants
  MCR (excluding PCR) | 21 | 14
  PCR | 29 | 11
  Nonclinical Response (NCR) | 119 | 63
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.4875, Wilcoxon (Mann-Whitney) — One-sided p-value

2. Secondary Outcome: Time-adjusted Area Under The Curve Minus Baseline (AUCMB) of BILAG Score Over The 52-week Treatment Period
Description: The BILAG Index measures clinical disease activity in SLE. A single alphabetic score (A through E) is used to denote disease severity for each of the 8 domains. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 8 domains. The AUCMB of BILAG Score Over 52 Weeks was calculated as: 1. Calculate the AUC of the BILAG global score versus time (in days) by 52 weeks. 2. Calculate the Time-Adjusted AUC by dividing the AUC by the number of days a patient was on the study. 3. Minus the Time-Adjusted AUC by the baseline BILAG global score
Time Frame: From baseline to 52 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: BILAG score unit
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 169 | 88
BILAG score unit | -5.8 (4.0) | -5.9 (4.5)
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.8230, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants Who Achieved an MCR (Excluding PCR)
Description: The BILAG Index measures clinical disease activity in SLE. A single alphabetic score (A through E) is used to denote disease severity for each of the 8 domains. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 8 domains. MCR = participants who achieved BILAG C scores or better at 24 weeks, maintained this response without developing a flare to 52 weeks, and did not experience a severe flare from Day 1 to Week 24. PCR = participants who achieved BILAG C score or better at 24 wks and maintained response without a flare for 16 consecutive weeks, or maximum of one BILAG B score at 24 weeks and maintained response without a flare to 52 wks, or maximum of 2 BILAG B scores at 24 wks without development of BILAG scores of A or B until Week 52 if the baseline BILAG score was 1A+>=2Bs, or>=2 As, or>=4 Bs, or participants who enrolled with scores of severe disease and did not achieve a single BILAG B at Month 6.
Time Frame: From baseline to 52 weeks
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 169 | 88
participants | 21 | 14
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.4318, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Participants Who Achieved a PCR (Including MCR)
Description: The BILAG Index measures clinical disease activity in SLE. A single alphabetic score (A through E) is used to denote disease severity for each of the 8 domains. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 8 domains. PCR = participants who achieved BILAG C score or better at 24 wks and maintained response without a flare for 16 consecutive weeks, or maximum of one BILAG B score at 24 weeks and maintained response without a flare to 52 wks, or maximum of 2 BILAG B scores at 24 wks without development of BILAG scores of A or B until Week 52 if the baseline BILAG score was 1A+>=2Bs, or>=2 As, or>=4 Bs, or participants who enrolled with scores of severe disease and did not achieve a single BILAG B at Month 6. MCR = participants who achieved BILAG C or better at 24 weeks, maintained this response without developing a flare to 52 weeks, and did not experience a severe flare from Day 1 to Week 24.
Time Frame: From baseline to 52 Weeks
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 169 | 88
participants | 50 | 25
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.9069, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants Who Achieved a BILAG C or Better in All Domains
Description: The BILAG Index measures clinical disease activity in SLE. A single alphabetic score (A through E) is used to denote disease severity for each of the 8 domains. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 8 domains.
Time Frame: 24 weeks
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 169 | 88
participants | 42 | 24
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.5602, Cochran-Mantel-Haenszel

6. Secondary Outcome: Time to First Moderate or Severe Flare
Description: The BILAG Index measures clinical disease activity in SLE. A single alphabetic score (A through E) is used to denote disease severity for each of the 8 domains. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 8 domains. A severe flare = participants had BILAG A score(s) present in one or more domains or BILAG B scores present in three or more domains at the same visit following a visit of inactive disease state defined above. A moderate flare = participants had only BILAG B scores present in two domains at the same visit following a visit of inactive disease state.
Time Frame: 52 weeks
Population: Number of participants who ever reached C/D/E for all 8 BILAG domains before Day 364 visit. If a participant reached C/D/E at the last visit, then this participant was excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 127 | 58
days | 112.0 [84.00 to 146.00] | 126.0 [56.00 to 225.00]
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.8979, Log Rank

7. Secondary Outcome: Change in SLE Expanded Health Survey Physical Function Score From Baseline
Description: Short Form (36) with additional questions specific to lupus (scale = 0-100; with 100 representing the highest level of functioning possible) to measure the ability of rituximab to improve quality of life. A positive value for this outcome measure indicates that symptoms have improved.
Time Frame: From baseline to 52 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 169 | 88
score on a scale | 8.2 (22.8) | 4.1 (17.9)
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.1277, ANCOVA

8. Secondary Outcome: Number of Participants Who Achieved an MCR in The ITT Population
Description: The BILAG Index measures clinical disease activity in SLE. A single alphabetic score (A through E) is used to denote disease severity for each of the 8 domains. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 8 domains. MCR = participants who achieved BILAG C scores or better at 24 weeks, maintained this response without developing a flare to 52 weeks, and did not experience a severe flare from Day 1 to Week 24.
Time Frame: From Weeks 24 to 52
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Number analyzed (Participants) | 169 | 88
participants | 14 | 9
Statistical Analysis 1: Comparison: Rituximab 1000 mg + Prednisone vs Placebo + Prednisone; Stratified by randomization factors (race and initial prednisone dose); Test type: Superiority or Other; p = 0.6202, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: From the beginning to the end of the study (Week 78 plus extended safety follow-up, with an average duration of 96 weeks).
Arm/Group | Rituximab 1000 mg + Prednisone | Placebo + Prednisone
Serious Adverse Events (participants affected / at risk) | 72/169 | 32/88
Other Adverse Events (participants affected / at risk) | 164/169 | 85/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg + Prednisone (N=169) | Placebo + Prednisone (N=88)
Neutropenia (Blood and lymphatic system disorders) | 6 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphophenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 2 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Diastolic Dysfunction (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 0 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Diverticular Perforation (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 1
Chest Pain (General disorders) | 2 | 3
Death (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Serum Sickness (Immune system disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 3
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 3
Bronchitis (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 0
Pneumonia Primary Atypical (Infections and infestations) | 1 | 0
Periorbital Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 1
Abdominal Abscess (Infections and infestations) | 0 | 1
Abscess Intestinal (Infections and infestations) | 1 | 0
Appendiceal Abscess (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3
Herpes Zoster (Infections and infestations) | 2 | 0
Herpes Virus Infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Gastroentiritis Viral (Infections and infestations) | 1 | 1
Cytomegalovirus Colitis (Infections and infestations) | 1 | 0
Genital Infection Female (Infections and infestations) | 0 | 1
Gastroentiritis Salmonella (Infections and infestations) | 0 | 1
Staphylococcal Bacteremia (Infections and infestations) | 0 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 1 | 1
Incision Hernia (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Drug Toxicity (Injury, poisoning and procedural complications) | 1 | 0
International Normalised Ratio Abnormal (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 3 | 4
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
SLE Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Spinal Cord Herniation (Nervous system disorders) | 1 | 0
Premature Labor (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Anxiety Disorder (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Lupus Nephritis (Renal and urinary disorders) | 3 | 3
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Abortion Induced (Surgical and medical procedures) | 1 | 2
Hypertension (Vascular disorders) | 2 | 1
Lupus Vasculitis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Febrile Infection (Infections and infestations) | 0 | 1
Disseminated Cytomegaloviral Infection (Infections and infestations) | 0 | 1
Viral Oesaphagitis (Infections and infestations) | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Mental Status Change (Psychiatric disorders) | 1 | 0
Hidradentis (Skin and subcutaneous tissue disorders) | 1 | 0
Venous Insufficiency (Vascular disorders) | 1 | 0
Substance-induced Psychotic Disorder (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg + Prednisone (N=169) | Placebo + Prednisone (N=88)
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Tachycardia (Cardiac disorders) | 10 | 3
Palpitations (Cardiac disorders) | 9 | 3
Cushingoid (Endocrine disorders) | 7 | 6
Vision Blurred (Eye disorders) | 3 | 5
Conjunctivitis (Eye disorders) | 4 | 6
Dry Eye (Eye disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 44 | 24
Vomiting (Gastrointestinal disorders) | 24 | 11
Diarrhoea (Gastrointestinal disorders) | 30 | 12
Abdominal Pain (Gastrointestinal disorders) | 12 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 12 | 5
Constipation (Gastrointestinal disorders) | 15 | 8
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 13 | 7
Abdominal Discomfort (Gastrointestinal disorders) | 10 | 5
Dyspepsia (Gastrointestinal disorders) | 8 | 7
Toothache (Gastrointestinal disorders) | 7 | 5
Oedema Peripheral (General disorders) | 25 | 13
Chest Pain (General disorders) | 10 | 9
Pain (General disorders) | 13 | 5
Fatigue (General disorders) | 21 | 15
Pyrexia (General disorders) | 17 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 54 | 32
Sinusitis (Infections and infestations) | 28 | 15
Nasopharyngitis (Infections and infestations) | 17 | 5
Urinary Tract Infection (Infections and infestations) | 48 | 26
Candidiasis (Infections and infestations) | 12 | 14
Oral Candidiasis (Infections and infestations) | 16 | 9
Bronchitis (Infections and infestations) | 28 | 12
Pneumonia (Infections and infestations) | 3 | 5
Herpes Zoster (Infections and infestations) | 16 | 4
Gastroenteritis Viral (Infections and infestations) | 9 | 7
Vulvovaginal Mycotic Infection (Infections and infestations) | 12 | 4
Gastroenteritis (Infections and infestations) | 15 | 2
Influenza (Infections and infestations) | 9 | 6
Ear Infection (Infections and infestations) | 2 | 5
Contusion (Injury, poisoning and procedural complications) | 10 | 6
Weight Increased (Investigations) | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 7
Decreased appetite (Metabolism and nutrition disorders) | 12 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 22 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 18 | 13
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 11 | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Joint Swelling (Musculoskeletal and connective tissue disorders) | 7 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 17 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 11 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 5
Headache (Nervous system disorders) | 38 | 23
Dizziness (Nervous system disorders) | 26 | 15
Migraine (Nervous system disorders) | 18 | 11
Hypoaesthesia (Nervous system disorders) | 8 | 5
Paraesthesia (Nervous system disorders) | 9 | 8
Insomnia (Psychiatric disorders) | 19 | 8
Anxiety (Psychiatric disorders) | 15 | 8
Depression (Psychiatric disorders) | 14 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 12
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Rash (Skin and subcutaneous tissue disorders) | 18 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 4
Erythema (Skin and subcutaneous tissue disorders) | 10 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 5
Hypertension (Vascular disorders) | 14 | 8
Flushing (Vascular disorders) | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.